CLINICAL TRIAL: NCT00367302
Title: Buprenorphine Maintenance for Opioid-Addicted Persons in Jail and Post-Release
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Western Michigan University (Other); New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Stephen Magura, Principal Investigator, Western Michigan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA020583; R21DA020583 (NIH); 1R21DA020583 (NIH)
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Opiate Addiction
Keywords: addiction; jail; opiates; buprenorphine; clinical trial
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Buprenorphine maintenance
  Interventions: Drug: buprenorphine
- 2 (Active Comparator): Methadone maintenance
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: buprenorphine — maintenance
  Other Names: Suboxone
  Arms: 1
Drug: methadone — maintenance
  Arms: 2

SUMMARY:
The purpose of the study is to determine the feasibility of providing buprenorphine maintenance to opioid-dependent offenders in a jail setting and of transitioning those patients to buprenorphine maintenance in the community after their release.

DETAILED DESCRIPTION:
Background: Heroin and other opioid abuse continues as a significant problem among the criminal justice population. In 2002, the criminal justice system was the source of referral for 36% of all substance abuse treatment admissions, the largest source of referrals. Heroin use among offenders has serious health and social consequences. Injection, still the primary route of administration among heroin users, is strongly associated with the transmission of HIV, hepatitis C and other blood-borne diseases. During 1997, 20% to 26% of all people living with HIV in the United States, and 29% to 43% of all those infected with hepatitis C, passed through a correctional facility. The relationship between heroin use and criminal activity has been extensively documented. Although methadone maintenance has been the primary treatment for chronic opioid dependence since the 1970's, correctional systems in the U.S., with very few exceptions (primarily Rikers Island in New York City), have not provided institutional access to methadone maintenance. Regrettably, negative attitudes to methadone are prevalent among criminal justice professionals, the public, treatment providers and opioid-dependent offenders themselves; there is little prospect of that changing soon. Buprenorphine maintenance is a recently approved therapy that may be more acceptable than methadone to the criminal justice system and opioid-dependent offenders. With one minor exception, buprenorphine has never been systematically administered as an opioid replacement therapy in a correctional setting in the U.S.

Aims and Objectives:

1. To determine the feasibility of providing buprenorphine maintenance to opioid-dependent offenders in a jail setting and of transitioning those patients to buprenorphine maintenance in the community after their release.
2. To conduct a randomized clinical trial of buprenorphine maintenance (N=50) vs. methadone maintenance (N=50) initiated in the jail setting and continuing in the community.
3. To determine the reasons that offenders fail to report for community buprenorphine or methadone treatment after release or drop out of community treatment.

Study Design: Consenting eligible inmates at Rikers Island in New York City will be randomly assigned to buprenorphine or methadone maintenance in jail and will be referred to a corresponding community treatment upon their release. Subjects will be followed-up at 3 months after release from jail.

Target Population: Opioid-dependent jail inmates sentenced to 10- 90 days.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependent patients who meet eligibility requirements for the KEEP program,
* patients serving sentences who will remain confined for at least 10 days but less than 90 days in the EMTC facility (all male) at Rikers,
* willingness to accept buprenorphine treatment,
* expected to reside in New York City after release
* 18-65 years of age

Exclusion Criteria:

* receiving methadone treatment in the community at sentencing and remanded to Rikers
* took non-prescribed 'street methadone' within last 3 days
* currently receiving more than 20mg/day methadone
* current psychotic symptoms (e.g., schizophrenia, schizoaffective disorder) requiring referral for mental health intervention, or current treatment with antipsychotic medication)
* HIV infection with T lymphocytes less than 200 per mm of blood and/or presence of a serious opportunistic infection requiring treatment, or receiving the HIV medication atazanavir.
* unable to complete English language interview

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Treatment completion in jail | Until release from jail
Reporting to assigned treatment modality after release | Within 3 months after release from jail

SECONDARY OUTCOMES:
Intention to continue treatment after release | At release from jail
Re-incarceration | Within 3 months after release
Frequency of illicit opioid use after release | Within 3 months after release
Re-arrest | Within 3 months after release
Severity of re-arrest charges | Within 3 months after release, if re-arrested
Satisfaction with opioid replacement treatment. | During jail and 3 months post-release
Opioid withdrawal symptoms and cravings | During jail and post-release

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Magura, Ph.D., Principal Investigator — Western Michigan University